CLINICAL TRIAL: NCT04525378
Title: Mesenchymal Stromal Cell-based Therapy for COVID-19-associated Acute Respiratory Distress Syndrome: a Pilot Clinical Study
Brief Title: MSC-based Therapy in COVID-19-associated Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCL02/2020
Record Dates: First submitted 2020-07-31; First posted 2020-08-25 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Covid19; ARDS, Human
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Patients will receive standard care.
- MSC - low dose (2.5x10ˆ7) (Experimental): Patients will receive standard care plus cell therapy.
  Interventions: Other: Mesenchymal stromal cell-based therapy
- MSC - intermediate dose (5x10ˆ7) (Experimental): Patients will receive standard care plus cell therapy.
  Interventions: Other: Mesenchymal stromal cell-based therapy
- MSC - high dose (10x10ˆ7) (Experimental): Patients will receive standard care plus cell therapy.
  Interventions: Other: Mesenchymal stromal cell-based therapy

INTERVENTIONS:
Other: Mesenchymal stromal cell-based therapy — Intravenous administration of MSCs, performed as single dose (high dose group) or repeated after 48 h (low doses; intermediate dose)
  Arms: MSC - high dose (10x10ˆ7); MSC - intermediate dose (5x10ˆ7); MSC - low dose (2.5x10ˆ7)

SUMMARY:
Considering the potential of mesenchymal stromal cells (MSCs) in the treatment of lung injuries by COVID-19, this pilot clinical trial evaluates the safety and potential efficacy of the cell therapy, administered intravenously, in patients with pneumonia associated with COVID-19-associated acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COVID-19 confirmed by RT-PCR;
* Thorax CT image suggestive of viral pneumonia;
* Respiratory failure (SaO2 <93% with O2 at 5L / min)
* Tracheal intubation (first 48 h);

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Patients with a history of cancer, chemotherapy in the past 2 years;
* Life expectancy less than 6 months or in exclusive palliative care;
* Severe liver failure, with Child-Pugh score> 12;
* High probability of death in the following 48 h;
* Previous renal failure: patients who were already on dialysis or patients with RFG <30ml / min / 1.73 m2;
* Clinical or radiological suspicion of tuberculosis and bacterial pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Intrahospital mortality | 28 days

SECONDARY OUTCOMES:
Length of stay in the ICU and Hospital | 28 days
Days without mechanical ventilation in 28 days | 28 days
PaO2 / FiO2 ratio | Day 1, Day 2 and Day 7 after cell infusion
Incidence of secondary infections | 28 days
Incidence of adverse events | 28 days
Quantification of inflammatory response markers | Day 1, Day 3 and Day 7 after cell infusion
  Exploratory evaluation of changes from baseline (percentage) in serum levels of CRP, LDH, Ferritin levels, a panel of cytokines, chemokines immune cell populations by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No